CLINICAL TRIAL: NCT03883204
Title: Neurocognitive Effectiveness in Treatment of First-episode Non-affective Psychosis: a Randomized Comparison of Aripiprazole and Risperidone Over 3 Years
Brief Title: Neurocognitive Effectiveness in Treatment of First-episode Non-affective Psychosis: 3-years Follow-up
Acronym: PAFIP3_nc3Y
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROAC2018_nc3Y
Record Dates: First submitted 2019-03-13; First posted 2019-03-20 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Psychotic Disorders; Psychosis
Keywords: Cognition; Antipsychotic Agents; Treatment; Effectiveness; Aripiprazole; Risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole (Active Comparator): Oral, dose range 10-30 mg/day, once or twice a day during study duration.
  Interventions: Drug: Aripiprazole
- Risperidone (Active Comparator): Oral, dose range 1-6 mg/day, once or twice a day during study duration.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Aripiprazole — Initial dose: 10 mg.
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Risperidone — Initial dose: 2 mg.
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
Cognitive enhancement is a primary goal in treating individuals with schizophrenia. Cognitive deficits are already present at the first break of the illness, seem to remain stable during early phases and noticeably influence daily functioning. Differences among antipsychotics in terms of cognitive effectiveness have turned out to be a topic of increasing research interest. The initially postulated superior neurocognitive effectiveness of second-generation antipsychotics (SGAs) compared to first-generation antipsychotics (FGAs) is currently under debate. Long-term studies would be of great value to evaluate the differential benefits exerted by antipsychotic drugs on cognitive performance. The aim of this study is to investigate the cognitive effects of aripiprazole and risperidone in first-episode psychosis at 3 years.

DETAILED DESCRIPTION:
Study setting and financial support: data for the present investigation were obtained from an ongoing epidemiological and three-year longitudinal intervention program of first-episode psychosis (PAFIP) conducted at the outpatient clinic and the inpatient unit at the University Hospital Marqués de Valdecilla, Spain. Conforming to international standards for research ethics, this program was approved by the local institutional review board. Patients meeting inclusion criteria and their families provided written informed consent to be included in the PAFIP. The Mental Health Services of Cantabria provided funding for implementing the program. No pharmaceutical company supplied any financial support.

Study design: this is a flexible-dose study of two neuroleptics (Aripiprazole and Risperidone) assigned at aleatory ratio 1:1. Rapid titration schedule (5-day), until optimal dose is reached, is a rule used unless severe side effects occur. At the treating physician's discretion, the dose and type of antipsychotic medication could be changed based on clinical efficacy and the profile of side effects during the follow-up period. Antimuscarinic medication, Lormetazepam and Clonazepam are allowed for clinical reasons. No antimuscarinic agents are administered prophylactically. Antidepressants (Sertraline) and mood stabilizers (lithium) are permitted if clinically needed.

Clinical assessment: the severity scale of the Clinical Global Impression (CGI) scale, the Brief Psychiatric Rating Scale (BPRS), the Scale for the Assessment of Positive symptoms (SAPS), the Scale for the Assessment of Negative symptoms (SANS), the Calgary Depression Scale for Schizophrenia (CDSS) and the Young Mania Rating Scale (YMRS) were used to evaluate symptomatology. To assess general adverse event experiences, the Scale of the Udvalg for Kliniske Undersogelser (UKU), the Simpson-Angus Rating Scale (SARS) and the Barnes Akathisia Scale (BAS) were used. The same trained psychiatrist (BC-F) completed all clinical assessments. These clinical data are described at AZQ2005 study.

Neuropsychological assessment. Cognitive functioning was assessed in patients at 2 points: baseline and 3 years after the initialization of antipsychotic treatment. The cognitive assessment at baseline was carried out at 12 weeks after recruitment because this time is considered optimal for patients' stabilization. The evaluation required approximately 2 h and was carried out in the same day by the same neuropsychologist (R.A.-A and E.G.-R). The neuropsychological battery comprises 9 cognitive domains: information processing speed, motor dexterity, working memory, verbal learning, visuospatial abilities, delayed memory, attention, executive function and theory of mind.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the First Episode Psychosis Clinical Program (PAFIP III) from January 2015 to December 2020.
* Experiencing their first episode of psychosis (First Episode of Psychosis is defined as that psychopathological state in which for the first time and regardless of its duration, the patient has enough severe psychotic symptoms to allow a diagnosis of psychosis, having received no specific psychiatric treatment for him).
* Living in the catchment area (Cantabria).
* No prior treatment with antipsychotic medication or, if previously treated, a total life time of adequate antipsychotic treatment of less than 6 weeks.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for brief psychotic disorder, schizophreniform disorder, schizophrenia, or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury with loss of consciousness.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Global cognitive index | 3 years
  In order to calculate a measure of Global Cognitive Functioning (GCF) raw cognitive scores were reversed when appropriate before standardization so they all have the same direction (the higher, the better). According to previous methodology, the GCF was calculated as T-scores, with raw scores of a healthy comparison sample. T scores were converted to deficit scores that reflect presence and severity of cognitive impairment. Deficit scores on all tests were then "averaged" to create the GCF score.

SECONDARY OUTCOMES:
Change in information processing speed | 3 years
  Measured by Wechsler Adult Intelligence Scale (WAIS)-III digit symbol subtest (standard total score).
Change in information processing speed | 3 years
  Measured by Trail Making Test (TMT) trail A.
Change in information processing speed | 3 years
  Measured by Continuoys Performace Test (CPT) reaction time.
Change in motor dexterity | 3 years
  Measured by Grooved Pegboard Test (time to complete with dominant hand).
Change in working memory | 3 years
  Measured by WAIS-III letter-number sequencing test (standard total score).
Change in working memory | 3 years
  Measured by WAIS-III digits forward (standard total score).
Change in verbal learning | 3 years
  Measured by the Rey Auditory Verbal Learning Test (RAVLT) (trials 1-5).
Change in visuospatial abilities | 3 years
  Measured by the Rey Complex Figure (RCF) (copy figure).
Change in delayed memory | 3 years
  Measured by the Rey Auditory Verbal Learning Test (RAVLT) (list recall and list recognition discrimination subscore).
Change in delayed memory | 3 years
  Measured by the Rey Complex Figure (RCF) (delayed recall).
Change in attention | 3 years
  Measured by Continuoys Performace Test (CPT) (discrimination subscores).
Change in executive function | 3 years
  Measured by Trail Making Test (TMT) trail B.
Change in executive function | 3 years
  Measured by Stroop Test (color-word).
Change in executive function | 3 years
  Measured by the Zoo Map Test (first and second conditions).
Change in executive function | 3 years
  Measured by the Tower of London Test (ToL) (total correct and total moves score).
Change in executive function | 3 years
  Measured by FAS Word Fluency and semantic (animal) fluency tests.
Change in theory of mind | 3 years
  Measured by Eyes Task (total correct score).

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Santander, Spain.
Locations (1):
- University Hospital Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No